CLINICAL TRIAL: NCT03439592
Title: Analysis of the Microbiota in Hyperglycemic and Normoglycemic Patients With ST Segment Elevation Myocardial Infarction (STEMI)
Brief Title: Analysis of the Microbiota and STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, assistant professor, University of Campania Luigi Vanvitelli
Other Study IDs: 142002018
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: STEMI; Diabetes Mellitus; Microbial Colonization
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Mellitus; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — we will collect fecal material obtained before, and during percutaneous coronary intervention in STEMI patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hyperglycemic patients: diabetic patients admitted for STEMI and with hyperglycemia at hospital admission.
  Interventions: Diagnostic Test: collection of fecal material
- normoglycemic patients: diabetic patients admitted for STEMI and with normoglycemia at hospital admission.
  Interventions: Diagnostic Test: collection of fecal material

INTERVENTIONS:
Diagnostic Test: collection of fecal material — in study population we will collect fecal material to analyze the microbiotic flora by genetic techniques.

SUMMARY:
Hyperglycemia is a common finding in patients diagnosed with acute coronary syndrome (ACS), and an independent predictor of mortality in patients with and without diabetes. Though percutaneous coronary intervention (PCI) is the cornerstone of ST-segment elevation myocardial infarction (STEMI), the incidence of heart failure, re-infarction and death in hyperglycemic patients remains significant, with a mortality of more than 40% one year after the event. In these STEMI patients dual anti-aggregation therapy is currently the gold standard after PCI, but bleeding phenomena, and therapeutic resistance may reduce their therapeutic efficacy. Therefore, it is likely that the individual response to the dual anti-aggregation therapy, and the hyperglycemic stress, may influence resistance mechanisms, and/or lead to an increase in pharmacological functional deactivation by the microbiotic flora. The term microbiota indicates the totality of the genomes of microorganisms that reside in an ecological niche, and which constitute the "human microbiota". In this context, the analysis of the faecal microbiota before PCI, at hospital discharge and at follow-up, could be considered useful for identifying hyperglycaemic patients with alteration of metabolic-oxidative processes, and pro-thrombotic correlates with worse post procedural prognosis. Therefore, the analysis of faecal microbiota during the STEMI event could theoretically identify hyperglycemic patients with excessive inflammatory and oxidative tone caused by hyperglycemia, conditioning resistance to double anti-aggregation therapy and coronary stenting, and conditioning pro-thrombotic phenomena after coronary reperfusion by PCI. Therefore, authors will conduct a study to analyze the microbiota in patients with acute hyperglycaemic and normoglycemic coronary syndrome. The primary objective of this study will be to evaluate any changes in the microbiota and its activity on faecal material taken before PCI, and after 6 and 12 months in patients with hyperglycemic STEMI, and also evaluate if the changes in the microbiota can be related to the 12-month prognosis.

DETAILED DESCRIPTION:
Hyperglycemia is a common finding in patients diagnosed with acute coronary syndrome (ACS) and is an independent predictor of mortality in patients with and without diabetes (1-4). Though percutaneous coronary intervention (PCI) is the cornerstone of ST-segment elevation myocardial infarction (STEMI) (4-6), the incidence of heart failure, re-infarction and death in hyperglycemic patients remains significant, with a mortality of more than 40% one year after the event (4-5). In fact, restenosis and no-reflow phenomena are common events leading to worse clinical outcomes, in hyperglycemic patients undergoing primary PCI, and resulting in atherothrombotic embolization, increased oxidative stress and inflammation (3-6). In an attempt to counter the increasing in mortality from hyperglycemia, the coronary units implemented insulin protocols to normalize blood glucose during ACS, and the same insulin treatment showed conflicting results (7). Data from small pilot studies, from moderate clinical trials and a meta-analysis suggested benefits from insulin therapy (1-3.5). On the other hand, subsequent randomized clinical trials have not confirmed an increase in survival (7, 8) . Moreover, if the dual anti-aggregation therapy is currently the therapeutic basis of patients with STEMI treated by PCI (9), increasingly frequent anti-aggregation therapy and bleeding phenomena, may reduce their therapeutic efficacy (11 -13). Therefore, it is likely that the individual response to the dual anti-aggregation therapy, and the hyperglycemic stress, may influence resistance mechanisms, and/or lead to an increase in pharmacological functional deactivation by the microbiotic flora. The term microbiota indicates the totality of the genomes of microorganisms that reside in an ecological niche, and which constitute the "human microbiota" (14). According to the analyzed anatomical district we speak of intestinal, ocular, buccal, vaginal microbiota, etc. The DNA analysis of microorganisms living in the human intestinal tract, realized with metagenomic methods by the MetaHIT consortium, has identified over 3 million genes, 150 times those of the human species (16-21). In addition, cardiovascular diseases such as hypertension and coronary artery disease are strongly conditioned by the presence of Enterobacteriaceae, Firmicutes and Lattobacilli in the intestine, which can determine their onset (22). In this context, the analysis of the faecal microbiota before PCI, at hospital discharge and at follow-up, could be considered useful for identifying hyperglycaemic patients with alteration of metabolic-oxidative processes, and pro-thrombotic correlates with worse post procedural prognosis ( 23). The ease of obtaining samples of faecal microbiota, and the relevant impact on the scientific community, and on routine clinical practice, pushes us to insist on clinical research, together with a genomic, metabolic and cellular analysis of the microbiota, and to extract as much information as possible in hyperglycemic patients with STEMI. This investigation has never been proposed in the scientific research and clinical practice of hospitalized hyperglycaemic patients for STEMI. Indeed, a large amount of evidence suggests that, hyperglycaemia causes an increasing production of oxidative stress and inflammation, both in atherosclerotic plaque and in the thrombus, and therefore it plays a central role in determining worse outcomes in STEMI. Therefore, the analysis of faecal microbiota during the event could theoretically identify hyperglycemic patients with excessive inflammatory and oxidative tone caused by hyperglycemia, conditioning resistance to double anti-aggregation therapy and coronary stenting, and conditioning pro-thrombotic phenomena after coronary reperfusion by PCI. Therefore, authors will conduct a study to analyze the microbiota in patients with acute hyperglycaemic and normoglycemic coronary syndrome.

OBJECTIVES The primary objective of this study will be to evaluate any changes in the microbiota and its activity on faecal material taken before PCI, and after 6 and 12 months in patients with hyperglycemic STEMI, and also evaluate if the changes in the microbiota can be related to the 12-month prognosis.

MATERIALS AND METHODS Patients This is a cohort study to investigate the effects of possible changes in the microbiota and its activity in faecal samples taken from patients with hyperglycemic STEMI v/s normoglycemic. These patients are treated according to routine "real life" therapeutic practices, adopted at the Cardiology Division of the "Luigi Vanvitelli" University of Campania. After discharge from the hospital, all patients will be invited to carry out the control visits, as indicated by the guidelines for the management of post-STEMI patients (6), at the Cardiology Division of the University of Campania "Luigi Vanvitelli "and at the VI Division of Internal Medicine of the" Luigi Vanvitelli "University of Campania. All patients will be monitored for 12 months after the event, as a follow-up. According to the recent definition of the American Heart Association, hyperglycemia will be defined by fasting blood glycemic levels> 140 mg / dl (1, 9). All patients with onset of symptoms within 12 hours and 1 mm elevation of the ST segment in 2 or more contiguous peripheral leads or at least 2 mm in 2 or more contiguous precordial leads or new onset left branch block will be considered for PCI. Inclusion criteria will include: age over 18 and admission for STEMI first episode. Patients with left ventricular ejection fraction <25%, with previous IMA or previous PCI and / or by-pass will be excluded. Each will be included in the study after signing an informed consent. Routine haematological analysis will be performed at the time of acceptance, before practicing medical therapy and possible coronary artery examination and after 6 and 12 months. On an aliquot of the blood sample taken at these times, we will evaluate trimethylamine-N-oxide (TMAO), a product of bacterial metabolism, whose elevated serum levels are associated with adverse cardiovascular events (24). In addition, before the PCI, and 6 and 12 months later, a stool sample will be taken on which the microbiota will be subsequently analyzed. The research will be conducted in accordance with the principles of the Helsinki declaration.

Procedure In this study authors will evaluate a cohort of patients with STEMI admitted to the Cardiology Division of the "Luigi Vanvitelli" University of Campania, and treated by dual anti-aggregating therapy. All patients will be treated according to the suggested protocols of the latest Guidelines on STEMI (6). Patients will be classified into two groups: hyperglycaemic patients v/s normoglycemic, in both groups of patients will be carried out analysis of the fecal microbiota, pre PCI and pre dual antiplatelet therapy. The microbiota will be extracted from faecal material, and then prepared and subsequently analyzed. It is not possible in clinical practice to culture in the laboratory the vast majority of intestinal bacteria, as compared to the enormous amount of microorganisms present. Thanks to the most up-to-date techniques of sequencing the bacterial DNA (Next Generation Sequencing) extracted from the faecal material, it is now possible a complete and reliable identification of the intestinal microbiota. In addition to identify the bacterial species present, authors are also able to express an overall health degree of the microbiota (or dysbiosis), its efficiency in the production of some useful or harmful substances, the adequacy of the microbiota with respect to some fundamental functions to which is a deputy and the propensity of the microbiota itself against inflammatory bowel diseases, metabolic diseases and aging. The result is an impressive amount of data, a true identity card of the microbiota, named the Microbiota passport.

Sample preparation and analysis. Samples for sequencing the microbiota will be collected from faecal material and stored at ultra-low temperature (-80°C) to avoid damage to the original sample. The sequencing of the microbiota will be performed by the laboratory of Microbiology of the University of Campania "Luigi Vanvitelli". For the sequencing of the microbiota we will use the "NextGeneration Sequencing" (NGS) method, which allows the sequencing in parallel of millions of DNA fragments (25) through the use of Illumina machinery (San Diego, CA). The DNA will be extracted from these samples using a high reproducibility commercial kit procedure (Qiagen, Invitrogen). The final yield and quality of the extracted DNA will be determined using the NanoDrop ND-1000 spectrophotometer (ThermoScientific, Waltham, MA) and QubitFluorometer 1.0 (Invitrogen Co., Carlsbad, CA). The extracted DNA will be amplified by PCR with the primers: forward: 5'-CCTACGGGNGGCWGCAG-3 'and reverse: 5'-GACTACHVGGGTATCTAATCC-3' (Klindworth et al.2013), which target the hypervariable region V3 and V4 of the 16S rRNA gene . Each PCR amplification will be performed by protocol for the preparation of 16S libraries for metagenomic sequencing (Illumina, San Diego, CA). The amplification products will be quantified by the Qubit fluoridator (Invitrogen Co., Carlsbad, CA) and grouped at an equimolar amount of each sample with a final concentration of 2nM. A Phix control library (Illumina) will be added to the samples. The grouped samples will then be sequenced on the MiSeq Platform (Illumina, San Diego, CA). The data thus obtained will be subjected to quality controls by bioinformatics analysis with FastQC. Finally, the data will be analyzed according to the statistical tests suggested by the guidelines for metagenomic sequencing. Patient data will be compared with each other and over time with reference databases. The evaluation of the epigenetic activity of the microbiota and the biochemical dosages of cytokines and free radicals will be performed at the laboratory of Pharmacology of the University of Campania "Luigi Vanvitelli. In particular, for the evaluation of the epigenetic activity of the microbiota of each individual hyperglycemic v/s normoglycemic patient with STEMI, we will proceed according to the protocol QIAGEN (Italy) with the extraction from faecal material of the total RNA, including the low-weight one molecular (microRNA). The final yield and quality of the extracted RNA will be determined using the NanoDrop ND-1000 spectrophotometer (ThermoScientific, Waltham, MA). Through qRT-PCR (QIAGEN, Italy) the expression levels of the following fecal microRNAs will be detected: miR-10b, miR-204, miR-29, miR-496, miR-1224-5p, miR-470 and miR-663 involved in the regulation of the intestinal microbiota; miR-10a and miR-18b involved in the regulation of intestinal microbiota and metabolic inflammation; miR-106a, miR-17, miR-19a, miR-20a, miR-206, miR-222 and miR-223 involved in metabolic inflammation and signaling insulin/IGF-1 (26). The metabolic activity of the microbiota in each individual hyperglycaemic v/s normoglycemic patient with STEMI will be evaluated by determination of short chain fatty acids (SCFA) from faecal samples: the levels of fecal SCFA, a product of bacterial fermentation, seem to correlate with an improvement in type 2 diabetes (27). The inflammatory activity of the microbiota will be evaluated by determining the fecal levels of LPS (28-29), IL-1β and IL-6 (30-32), while the oxidative activity through the analysis of fecal levels of ROS, SOD and GSH (33-34).

Follow-up Authors' study is designed to manage hyperglycaemic v/s normoglycemic patients with STEMI in the "real life", without interference from the rigid rules that limit the generalisability of RCTs. Therefore, after discharge from the hospital, all patients will be invited to carry out the control visits, as indicated by the guidelines for the management of post-STEMI patients (6), at the Cardiology Division of the University of Campania "Luigi Vanvitelli", and at the VI Division of Internal Medicine of the "Luigi Vanvitelli" University of Campania. All patients will be monitored for 12 months after the event, as follow-up, to practice clinical evaluation (ECG, exercise test, echocardiogram, glucose levels), as indicated by the guidelines for the management of STEMI patients (6). At these time points, stool samples will also be taken for the analysis of the microbiota. Moreover, in the management and assessment of the glycemic compensation in the 12 months of follow-up, the physician will also be involved in order to maintain HbA1c levels <7%, glycemia between 90 and 140 mg / dl and postprandial glycemia <180 mg / dl.

Cardiovascular endpoints The cardiovascular end points in both cohorts will include myocardial re-infarction, re-hospitalization for coronary artery disease (re-stenosis, stent implantation or aorto-coronary bypass), heart failure, stroke, cardiac mortality, and all causes of mortality. The primary composite end point will consist of cardiovascular events, such as myocardial infarction, hospitalization for heart failure, stroke or cardiac mortality. The secondary end point will consist in the evaluation of cardiac function: reduction of ejection fraction, increase in volume of the left ventricle, reduction of coronary perfusion. All deaths will be reviewed and classified as cardiac (death caused by IMA, ventricular arrhythmias, refractory heart failure) or non-cardiac. All revascularizations will be classified as early (elective revascularization within 60 days after coronary angiography) or late. Only late revascularizations will be classified as cardiac events, so patients with early elective revascularization will be excluded from the analysis.

Statistical analysis The two groups will be compared using the Pearson χ2 test for categorical variables and the Kruskal-Wallis test for continuous variables. The covariate candidates for entry into the multivariable model will be identified by concentrating on the factors those that will significantly differ (P value <0.05) in the univariate analysis between hyperglycemic v/s normoglycemic patients. Cox regression will be used to build the mortality model. The Hazard Ratio for mortality will be adjusted for age, BMI, cholesterol, LDL, triglycerides and aspirin therapy, ticlopidine, combination of anti-aggregants, β-blockers, ACE inhibitors or sartans, antidiabetics, statins, during hospitalization for STEMI. Survival analysis through the first year from STEMI will be performed using the Kaplan-Meier curve and Cox regression method. The mortality curves will be obtained separately for hyperglycaemic patients v/s normoglycemia, to be compared using the log-rank test. All tests will be considered significant if p value <0.05. All analyzes will be carried out in the two study populations. A "propensity score" analysis will be performed using a "non parsimonious" logistic regression model that will compare the outcomes of the hyperglycemic v / s normoglycemic patients. More variables will be included in the model including age, sex, diabetes, hypertension, hypercholesterolemia, multivessel disease, chronic renal failure, TIMI pre-procedure flow, ejection fraction and procedural success. The C-score will indicate good discrimination. Based on the "matched" samples, the Cox proportional risk model will be used to determine the impact of hyperglycemia, and of microbiotic flora activity on mortality during follow-up. SPSS (version 21, IBM SPSS) will be used for all analyzes.

Sample Size The Sample Size will be calculated with IBM PC computer by GPOWER software. The size effect will be calculated according to the epidemiological and interventional studies performed on hyperglycaemic patients. The sample size estimated on a global effect of 25% with type I error of 0.05 and a power of 95% will be 200 participants, 100 for the group composed of normoglycemic patients and 100 for the group of hyperglycaemic patients.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years
* STEMI acute admission event

Exclusion Criteria:

* left ventricular ejection fraction <25%,
* previous acute myocardial infarction
* previous percutaneous coronary intervention
* previous coronary artery by-pass

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with hyperglycemic STEMI v/s normoglycemic STEMI. All patients with onset of symptoms within 12 hours and 1 mm elevation of the ST segment in 2 or more contiguous peripheral leads or at least 2 mm in 2 or more contiguous precordial leads or new onset left branch block will be considered for percutaneous coronary intervention (PCI). Patients aged over 18 and admitted for first STEMI episode.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
all cause deaths | 12 months
  authors will evaluate form hospital discharge schedules, and during follow up by clinical visits the deaths events for all causes.
cardiac deaths | 12 months
  authors will evaluate form hospital discharge schedules, and during follow up by clinical visits the deaths events for cardiac causes.

CONTACTS AND LOCATIONS:
Overall Officials: raffaele marfella, MD, PhD, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deedwania P, Kosiborod M, Barrett E, Ceriello A, Isley W, Mazzone T, Raskin P; American Heart Association Diabetes Committee of the Council on Nutrition, Physical Activity, and Metabolism. Hyperglycemia and acute coronary syndrome: a scientific statement from the American Heart Association Diabetes Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2008 Mar 25;117(12):1610-9. doi: 10.1161/CIRCULATIONAHA.107.188629. Epub 2008 Feb 25. PMID 18299505
- [Derived] Sardu C, Consiglia Trotta M, Santella B, D'Onofrio N, Barbieri M, Rizzo MR, Sasso FC, Scisciola L, Turriziani F, Torella M, Portoghese M, Loreni F, Mureddu S, Lepore MA, Galdiero M, Franci G, Folliero V, Petrillo A, Boatti L, Minicucci F, Mauro C, Calabro P, Feo M, Balestrieri ML, Ercolini D, D'Amico M, Paolisso G, Galdiero M, Marfella R. Microbiota thrombus colonization may influence athero-thrombosis in hyperglycemic patients with ST segment elevation myocardialinfarction (STEMI). Marianella study. Diabetes Res Clin Pract. 2021 Mar;173:108670. doi: 10.1016/j.diabres.2021.108670. Epub 2021 Jan 14. PMID 33453294
- [Derived] Sardu C, Pieretti G, D'Onofrio N, Ciccarelli F, Paolisso P, Passavanti MB, Marfella R, Cioffi M, Mone P, Dalise AM, Ferraraccio F, Panarese I, Gambardella A, Passariello N, Rizzo MR, Balestrieri ML, Nicoletti G, Barbieri M. Inflammatory Cytokines and SIRT1 Levels in Subcutaneous Abdominal Fat: Relationship With Cardiac Performance in Overweight Pre-diabetics Patients. Front Physiol. 2018 Aug 21;9:1030. doi: 10.3389/fphys.2018.01030. eCollection 2018. PMID 30246793